CLINICAL TRIAL: NCT05486910
Title: Evaluation of the Management of Side-Effects of Anti-Acne Treatment by a Cosmetic Routine Following Failure of the Usual Cosmetic Routine
Brief Title: Management of Side-Effects of Anti-Acne Treatment by a Cosmetic Routine
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: LRP20026-EFFACLAR SENSIBIOME
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Acne
Keywords: acne; efficacy; tolerance; dermocosmetic; quality of life
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retinoid-based topical acne treatment may induce local tolerance issues such as erythema, dryness, stinging and burning sensations that may reduce adherence and efficacy.

The tested regimen (cream and cleanser) has been specifically developed to rebalance the skin microbiome and compensate side-effects of topical treatments (hydration, skin barrier repair) together with an action on skin imperfections and marks.

This open-label study was conducted in subjects aged 12 years and over with sensitive skin (>2 on a sensitivity composite score from 0-3) treated for at least one month with the fixed-dose gel combination and presenting with treatment-related skin intolerance.

DETAILED DESCRIPTION:
The study on the evaluation of the management of side-effects of an anti-acne treatment by a cosmetic routine (cleanser and cream) following failure of the usual cosmetic routine has been conducted under dermatological control by Dermscan that is certified by the International Standards Organization (ISO) 9001-2015.

Each study report is subjected to a quality inspection by a proofreader member of Dermscan not involved in the audited study. The inspection of the study report allows to confirm that the results reflect exactly the study raw data and that the study fulfills any standard and regulatory requirements.

Regarding the statistical analysis, data obtained for each parameter, at each measurement time and on each zone are presented in raw value tables. The tables also show the descriptive statistics: means, medians, minima, maxima, standard errors of the means (SEM), confidence intervals of 95% (CI 95%) of these values as well as the variations and percentage variations. They also present the results of the statistical analysis.

Participants have the right to exit from the study at any time and for any motive in compliance with the Helsinki Declaration (1964) and its successive updates. The investigator can also interrupt the subject participation in the study prematurely in the case of a disease occurrence, a pregnancy or the occurrence of an adverse reaction.

The personnel in charge of the study collects data into individual case report forms in electronic or paper format and/or directly from measurement software. When information is collected in paper format, the double data entry is then done from these supports by the designed operator(s), without any interpretation, in specific EXCEL databases. The Project Manager or assistant checks the double data entry by comparing both databases. Then the coherence of the whole data set is checked as well as formulas used in the EXCEL tables (calculation formulas, selected data…). When all the controls are done, the database is locked.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian;
* phototype I to IV
* subject under EPIDUO® with a failed cosmetic routine for more than 1 month.
* subject agreeing to change their routine (introduction of the EFFACLAR routine).
* subjects with moderate skin sensitivity: composite score >2 at the inclusion (burning sensation, tightness and itching) with 4 grades: absent, slight, medium and severe
* subject under anti-acne treatment since 1 month, with an usual routine in failure
* subject who presents irritated skin due to EPIDUO® treatment

Exclusion Criteria:

* pregnant or nursing woman or woman planning a pregnancy during the study
* cutaneous pathology on the studied zone other than acne (eczema etc.)

  • use of topical or systemic treatment during the previous weeks liable to interfere with the assessment of the cutaneous acceptability of the study product (according to the investigator's appreciation, except the anti-acne treatment Epiduo and former cosmetic routine)
* oral treatment of retinoids during the six previous months of the study
* any change in hormonal treatment (including contraceptive) during the three previous months of the study or subject under Androcur® generic) treatments since less than six months
* professional facial care during the study or within the previous month
* subject manipulating her/ his acne lesions
* excessive exposure to sunlight or UV-rays within the previous month

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: participants with a failed anti-acne routine meeting the inclusion and exclusion criteria and agreeing to the study constraints
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
change in comedogenic potential | from baseline to Day28
  counting of retentional and inflammatory elements on the whole face. Descriptive statistics are done in order to determine the variation significance.
change in Global Evaluation Acne (GEA) score | from baseline to Day28
  The dermatologist realizes clinical score on the face using the Investigator Global Acne Severity Score : from 0 Clear. No lesions to 5 Very severe.

SECONDARY OUTCOMES:
change in sensitivity score by the dermatologist | from baseline to Day28
  evaluation of the parameters erythema, dryness, desquamation on a 0-3 scale
change in sensitivity score by the participant (composite score) | from baseline to Day28
  evaluation of the parameters itching, tightness, burning sensation on a 0-3 scale
change in global tolerance score by the dermatologist | from baseline to Day28
  evaluation of the tolerance on a 0-3 scale
change in global tolerance score by the participant | from baseline to Day28
  evaluation of the tolerance on a 0-3 scale
change in overall effectiveness score by the dermatologist | from baseline to Day28
  evaluation of the effectiveness on a 0-3 scale
change in overall effectiveness score by the participant | from baseline to Day28
  evaluation of the effectiveness on a 0-3 scale
change in quality of life | from baseline to Day28
  Cardiff Acne Disability Index (CADI) questionnaire with 5 questions

CONTACTS AND LOCATIONS:
Overall Officials: Anna Czermanska, Study Director — Eurofins
Locations (1):
- Studio Dermatologia i Kosmetyka, Malbork, Poland